CLINICAL TRIAL: NCT06331962
Title: The Effects of Remote Exercise Program in Patients With Digestive Tract Cancer and Chemotherapy-induced Peripheral Neuropathy
Brief Title: Digestive Tract Cancer and CIPN
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Cheng-Kung University Hospital (Other)
Collaborators: National Cheng Kung University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B-ER-112-010
Record Dates: First submitted 2023-12-11; First posted 2024-03-26 (Actual); Last update posted 2024-03-26 (Actual); Status verified 2023-08

CONDITIONS: Digestive Tract Cancer; Chemotherapy-induced Peripheral Neuropathy; Remote Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- remote home-based exercise therapy group (Experimental): Location and Frequency: Four times per week at the individual's own home. Exercise Duration: Eight weeks (subject to adjustments based on actual progress), with a total exercise time of 40 minutes each session.
  Exercise Components: Cardiovascular endurance exercise, resistance training, sensory exercises.
  Note: The participant will receive a customized exercise plan based on their capabilities, including guidelines and exercise instructions (exercise names, required equipment, movement sequences, repetitions, precautions).
  Interventions: Other: remote home-based exercise therapy group
- supervised exercise therapy group (Active Comparator): Exercise Location and Frequency: Physiotherapy Center (twice a week) and individual's home (twice a week).
  Exercise Duration: Eight weeks (subject to adjustments based on actual progress), with a total exercise time of 40 minutes each session.
  Exercise Components: Cardiovascular endurance exercise, resistance training, sensory training exercises. The home-based exercise training content is partially the same as the remote home-based exercise group.
  Interventions: Other: supervised exercise therapy group
- regular care group (Other): Perform regular care for eight consecutive weeks. After the tracking period ends (8 weeks), provide home-based education on resistance exercises, cardiovascular endurance exercises, and sensory training exercises.
  Interventions: Other: regular care group

INTERVENTIONS:
Other: remote home-based exercise therapy group — Location and Frequency: Four times per week at the individual's ownhome. Exercise Duration: Eight weeks (subject to adjustments based onactual progress), with a total exercise time of 40 minutes each session.
  Exercise Components: Cardiovascular endurance exercise, resistancetraining, sensory exercises.
  Note: The participant will receive a customized exercise plan based ontheir capabilities, including guidelines and exercise instructions (exercisenames, required equipment, movement sequences, repetitions,precautions).
  Arms: remote home-based exercise therapy group
Other: supervised exercise therapy group — Exercise Location and Frequency: Physiotherapy Center (twice a week)and individual's home (twice a week).
  Exercise Duration: Eight weeks (subject to adjustments based on actualprogress), with a total exercise time of 40 minutes each session.
  Exercise Components: Cardiovascular endurance exercise, resistancetraining, sensory training exercises. The home-based exercise trainingcontent is partially the same as the remote home-based exercise group.
  Arms: supervised exercise therapy group
Other: regular care group — Perform regular care for eight consecutive weeks. After the trackingperiod ends (8 weeks), provide home-based education on resistanceexercises, cardiovascular endurance exercises, and sensory trainingexercises.
  Arms: regular care group

SUMMARY:
According to the incidence rate of cancer, the digestive tract cancer accounts for two of the top ten cancers. It also accounts for half of the top ten causes of cancer death. Chemotherapy remains one of the most common forms of cancer treatment, and chemotherapy-induced peripheral neuropathy (CIPN) is one of the common adverse effects of cancer treatment in cancer survivors. To date, there is no exercise guideline established for patients with CIPN; therefore, CIPN remains quite threatening to cancer survivors. Due to limited studies on effects of exercise on improvement of CIPN symptoms in patients with digestive tract cancers, this study aims to investigate the effects of exercise and different intervention delivery modes (remote home exercise and exercise under supervision) at different time points on the CIPN symptoms, body inflammatory index, physical function, and quality of life of gastrointestinal cancer survivors with chemotherapy-induced peripheral neuropathy.

ELIGIBILITY:
Inclusion Criteria:

1. Age 20 and above;
2. Diagnosed by a physician with gastrointestinal cancer and has undergone chemotherapy or is currently undergoing chemotherapy;
3. Diagnosed by a physician with chemotherapy-induced peripheral neuropathy.

Exclusion Criteria:

1. Cognitive impairment or inability to cooperate with verbal instructions;
2. Neurological, muscular, skeletal, or cardiovascular issues preventing participation in exercise training;
3. Age 80 or above;
4. Refusal to engage in exercise intervention or participate in data collection.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2023-05-19 (Actual); Primary Completion 2025-07-31 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
Basic information | baseline, 4-week intervention, 8-week intervention, and 3 month after intervention
  Gender, date of birth, education level, survival days and status, exercise habit, alcohol consume history, smoking history, type of cancer, stage of cancer, start date of chemotherapy, number of chemotherapy sessions prior to intervention, chemotherapy drugs used, study period, and the subjects' medical history.
gene | baseline
  gene
body height | baseline, 4-week intervention, 8-week intervention, and 3 month after intervention
  body height in m
body weight | baseline, 4-week intervention, 8-week intervention, and 3 month after intervention
  body weight in kg
body mass index | baseline, 4-week intervention, 8-week intervention, and 3 month after intervention
  body mass index in kg/m2
blood data | baseline, 4-week intervention, 8-week intervention, and 3 month after intervention
  blood data, including blood cell count, neutrophils, lymphocytes, monocytes, hemoglobin, albumin, magnesium, mean corpuscular volume, etc.
Questionnaire of Quality of Life | baseline, 4-week intervention, 8-week intervention, and 3 month after intervention
  The European Organization for Research and Treatment of Cancer Quality of Life Questionnaire-Core 30 (QLQ-C30) is to assess the quality of life. The transferred score range for this tool is typically from 0 to 100, where 0 indicates very poor quality of life, and 100 indicates very good quality of life. There are five aspects in the QLQ-C30, including physical functioning, role functioning, emotional functioning, cognitive functioning, and social functioning. In this scoring system, higher scores generally indicate better quality of life, while lower scores suggest poorer quality of life.
Questionnaire of Chemotherapy-Induced Peripheral Neuropathy | baseline, 4-week intervention, 8-week intervention, and 3 month after intervention
  The European Organisation for Research and Treatment of Cancer Chemotherapy-Induced Peripheral Neuropathy 20-item scale (CIPN-20) assesses sensory abnormalities in patients. Scores range from 0 to 80, with 0 indicating no abnormalities and 80 severe abnormalities. Lower scores indicate better outcomes, while higher scores indicate worse outcomes. The total score is calculated by adding scores from items 1 to 19, ranging from 19 to 76, termed the CIPN20 sum1-19 score. Item 20 evaluates male impotence, relevant only for males. Additionally, items are categorized into sensory (1, 2, 3, 4, 5, 6, 9, 10, and 18), motor (7, 8, 11, 12, 13, 14, 15, and 19), and autonomic (16, 17, and 20) subscales.

SECONDARY OUTCOMES:
Muscle Strength | baseline, 4-week intervention, 8-week intervention, and 3 month after intervention
  Evaluate muscle strength using grip strength assessment device. Participant grips device withdominant hand using maximum effort.
Dynamic Balance | baseline, 4-week intervention, 8-week intervention, and 3 month after intervention
  Use Timed Up & Go (TUG) test. Participant stands from chair upon signal, walks 3m at normal pace,returns, and sits. Time recorded
Sensation Test | baseline, 4-week intervention, 8-week intervention, and 3 month after intervention
  Assess sensory issues from neuropathy using Romberg test
Cardiovascular Endurance | baseline, 4-week intervention, 8-week intervention, and 3 month after intervention
  Assess using 2-min step test. Participant steps in place for 2 mins, feet higher thanmidpoint between patella and iliac spine. Tester notes successful steps in 2 mins.

CONTACTS AND LOCATIONS:
Overall Officials: Cheng-Feng Lin, Ph.D, Study Chair — Department of Physical Therapy, National Cheng-Kung University
Locations (1):
- Department of Physical Therapy, National Cheng-Kung University, Tainan, Taiwan